CLINICAL TRIAL: NCT01107587
Title: Reactogenicity and Safety of Two Doses of GlaxoSmithKline (GSK) Biologicals' Oral Live Attenuated Liquid Human Rotavirus (HRV) Vaccine 444563, in Healthy Infants
Brief Title: Study to Assess the Safety of GSK Biologicals' Liquid Human Rotavirus Vaccine in Healthy Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 113518
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Infections, Rotavirus
Keywords: Human rotavirus vaccine
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- HRV group (Experimental): Subjects will receive GSK Biologicals' human rotavirus vaccine 444563.
  Interventions: Biological: GSK Biologicals' human rotavirus vaccine 444563
- Placebo Group (Placebo Comparator): Subjects will receive placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GSK Biologicals' human rotavirus vaccine 444563 — Oral, two doses.
  Arms: HRV group
Biological: Placebo — Oral, two doses.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to assess the reactogenicity and safety of GSK Biologicals' liquid human rotavirus vaccine in healthy infants aged 6 to 16 weeks at the time of the first dose of vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) can and will comply with the requirements of the protocol.
* A male or female infant of Chinese origin between, and including, 6 and 16 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/ Legally Acceptable Representative(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of 36 to 42 weeks inclusive.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth (for corticosteroids, this will mean prednisone, or equivalent, >= 0.5 mg/kg/day. Inhaled and topical steroids are allowed).
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of the human rotavirus vaccine or placebo except for the routine childhood vaccinations.
* Any clinically significant history of gastrointestinal disease including any uncorrected congenital malformation of the gastrointestinal tract that would predispose for intussusception.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment..
* History of confirmed rotavirus gastroenteritis.
* Gastroenteritis within 7 days preceding the study vaccine or placebo administration.
* Previous vaccination with rotavirus vaccine or planned to use during the study period.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.

Ages: 6 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2010-04-13 (Actual); Primary Completion 2010-06-28 (Actual); Study Completion 2010-06-28 (Actual)

PRIMARY OUTCOMES:
Occurrence of grade 3 solicited adverse events. | Within the 8-day (Day 0 - 7) follow-up period after each vaccine dose.

SECONDARY OUTCOMES:
Occurrence of each solicited adverse event. | Within the 8-day (Day 0 - 7) follow-up period after each vaccine dose.
Occurrence of unsolicited adverse events. | Within the 31-day (Day 0 - 30) follow-up period after any vaccine dose.
Occurrence of serious adverse events. | Throughout the study period (Day 0 to Month 2).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Liucheng County, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Li RC, Li YP, Mo ZJ, Luo D, Huang T, Kong JL, Wang LH, Song NS, Liu A, Zhang H, Liao X, Karkada N, Han HH. Reactogenicity and safety of a liquid human rotavirus vaccine (RIX4414) in healthy adults, children and infants in China: randomized, double-blind, placebo-controlled Phase I studies. Hum Vaccin Immunother. 2013 Aug;9(8):1638-42. doi: 10.4161/hv.25076. Epub 2013 Jun 4. PMID 23807360
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113518 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/113518?search=study&b%22b''%22#rs
- Available data/document: Dataset Specification: 113518 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113518 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113518 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113518 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113518 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113518 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register